CLINICAL TRIAL: NCT07049406
Title: The Role of Cultural Beliefs on Eye Health Practices Across Communities in District Rahim Yar Khan
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/917
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Eye Strain
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Structured Pre-tested — This will analyzed forthe differences in cultural perceptions and their Influence on health-seeking behavior.

SUMMARY:
This study explores the role of cultural beliefs on eye health practices across communities in District Rahim Yar Khan, employing a mixed-methods approach to gather both quantitative and qualitative data. The research aims to identify the cultural beliefs and practices that influence eye health behaviors and outcomes in the region.

DETAILED DESCRIPTION:
Through surveys, interviews, and focus groups with community members, eye care professionals, and traditional healers, the study will provide insights into the complex relationships between cultural beliefs and eye health. The findings will inform the development of culturally sensitive eye health interventions and programs, ultimately contributing to improved eye health outcomes in the region.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18+ of any gender
* Have experienced eye health issues, and express awareness of or adherence to cultural beliefs related to health.

Exclusion Criteria:

* Individuals with significant cognitive impairments or language barriers
* Other Ocular disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study explores the role of cultural beliefs on eye health practices across communities in District Rahim Yar Khan, employing a mixed-methods approach to gather both quantitative and qualitative data. The research aims to identify the cultural beliefs and practices that influence eye health behaviors
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pre-designed performa | 12 Months
  eye health related and clututal belief catorigal quesioners

CONTACTS AND LOCATIONS:
Locations (1):
- hospitals in RYK, Rahim Yar Khan, Pakistan

IPD SHARING:
Plan to Share IPD: No